Version 1.3 28.1.2024

## CONSENT TO PARTICIPATE TO THE STUDY

Neutralized local anaesthesia versus non-neutralized local anaesthesia in the surgical treatment of carpal tunnel syndrome. A double-blinded, randomized controlled trial.

Kuopio University Hospital, Orthopaedics, traumatology and Hand Surgery Unit.

| \_\_\_\_\_\_ have been asked to participate in the above-mentioned scientific study, the purpose of which is to evaluate the effect of neutralizing local anaesthetic, i.e. changing the acidity of the solution closer to the acidity of the body, on the pain experienced during injection of local anaesthetic.

I have read and understood the written research information I received. From the release, I have received a sufficient explanation of the research and the collection, processing and disclosure of personal data to be carried out in connection with it. The contents of the release have also been told to me verbally, I have had the opportunity to ask questions and I have received sufficient answers to all my questions regarding the research.

I have had sufficient time to consider my participation in the study. I have received sufficient information about my rights, the purpose of the research and its implementation, as well as the benefits and risks of the research. I have not been pressured or enticed to participate in the study.

The information was provided by / / 20 .

I know that my information will be treated confidentially and will not be disclosed to third parties. (If data is disclosed, an explanation of who the data collected during the research can be disclosed to and how the confidentiality of the data is protected. If the research involves international cooperation, a separate data disclosure section should be added to the consent).

I understand that my participation is voluntary. I understand that I can withdraw this consent at any time without giving a reason and my withdrawal will not change the treatment I receive will in any way.

I am aware that if I interrupt the research or withdraw consent, the data collected from me up to the time of interruption and withdrawal of consent can be used as part of the research material.

Version 1.3 28.1.2024 2

| With my signature, I confirm my participation in this study and voluntarily | / |
|---|---|
| agree to be a research subject. | |

| Subject's name | Subject's date of birth | Address of the subject |
|---|---|---|
| Date | Signature | |
| Consent received | | |
| Name of study physica<br>(Consent recipient) | an/nurse Date | Signature |

The original signed consent of the research subject and a copy of the research information remain in the research doctor's archive. The study information sheet and a copy of the signed consent are given to the subject.